CLINICAL TRIAL: NCT01021332
Title: An Open-label, Long Term, Multi-center Study to Assess the Safety and Efficacy of Fixed Dose Combinations of Solifenacin Succinate (6 mg and 9 mg) With Tamsulosin Hydrochloride OCAS 0.4 mg, in Male Subjects With Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH) With a Substantial Storage Component
Brief Title: Long Term Study of Solifenacin Succinate and Tamsulosin Hydrochloride Oral Controlled Absorption System (OCAS) in Males With Lower Urinary Tract Symptoms
Acronym: Neptune II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-CL-057; 2008-001212-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Vesomni; Solifenacin succinate; EC905; Tamsulosin hydrochloride OCAS; Treatment; Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total Group (Experimental): Participants who received at least one dose of open-label fixed dose combination (FDC) treatment
  Interventions: Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/6 mg); Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/9 mg)

INTERVENTIONS:
Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/6 mg) — oral
  Other Names: EC905; Vesomni
Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/9 mg) — oral
  Other Names: EC905

SUMMARY:
Clinical study to examine the safety, tolerability and efficacy of long-term combination therapy of tamsulosin and solifenacin in the treatment of males with lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH) with a substantial storage component.

DETAILED DESCRIPTION:
This is an open-label extension study following the double blind 905-CL-055 study

ELIGIBILITY:
Inclusion Criteria:

* Completion of 12 weeks double-blind treatment in Study 905-CL-055

Exclusion Criteria:

* Any significant PVR volume (>150 mL)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2010-04-26 (Actual); Primary Completion 2011-12-14 (Actual); Study Completion 2011-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Global Development
Locations (66):
- Austria (2):
  - Innsbruck
  - Vienna
- Minsk, Belarus
- Belgium (5):
  - Antwerp
  - Edegem
  - Ghent
  - Leuven
  - Liège
- Czechia (7):
  - Hradec Králové
  - Ostrava
  - Pilsen
  - Roudnice nad Labem
  - Uherské Hradiště
  - Ústí nad Labem
  - Zd'ar Nad Sazavou
- France (5):
  - Colmar
  - Montluçon
  - Orléans
  - Paris
  - Pierre-Bénite
- Germany (16):
  - Bautzen
  - Eisleben Lutherstadt
  - Frankfurt
  - Ganderkesee
  - Hagenow
  - Halle
  - Hamburg
  - Henningsdorf
  - Hettstedt
  - Koblenz
  - Leipzig
  - Neustadt in Sachsen
  - Radebeul
  - Sachsen
  - Trier
  - Uetersen
- Italy (4):
  - Avellino
  - Catanzaro
  - Palermo
  - Treviglio
- Netherlands (7):
  - Amsterdam
  - Apeldoorn
  - Doetinchem
  - Maastricht
  - Sneek
  - Tilburg
  - Winterswijk
- Poland (6):
  - Bielsko-Biala
  - Bydgoszcz
  - Krakow
  - Puławy
  - Warsaw
  - Więcbork
- Slovakia (5):
  - Nitra
  - Piešťany
  - Prešov
  - Skalica
  - Trenčín
- United Kingdom (8):
  - Cardiff
  - Chorley
  - Liverpool
  - Northwood
  - Oxford
  - Reading
  - Sheffield
  - Taunton

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=39

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible for Study 905-CL-057 if they completed 12 weeks of double-blind treatment in Study 905-CL-055, complied with inclusion criteria and did not meet any exclusion criteria. Participants treated with the FDC 0.4 mg/6 mg or 0.4 mg/9 mg for maximally 40 weeks.
Pre-assignment Details: All eligible participants started with 4 weeks of open-label FDC 0.4 mg/6 mg and were given the opportunity to adjust their dose at 3 monthly intervals thereafter if desired.
Groups:
- Total Group: Participants who received at least one dose of open-label FDC treatment
Period: Overall Study
Arm/Group | Total Group
Started | 1066 (Took ≥ 1 dose of FDC open-label study drug)
Safety Analysis Set (SAF) | 1066
Full Analysis Set (FAS) | 1009
Completed | 960
Not Completed | 106
Not completed — Not fulfilling incl./excl.criteria | 5
Not completed — Adverse Event | 43
Not completed — Lack of Efficacy | 19
Not completed — Withdrawal of Consent | 23
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 9
Not completed — Miscellaneous | 3

BASELINE CHARACTERISTICS:
Population: SAF and FAS (study-specific)
Arm/Group | Total Group
Number analyzed (Participants) | 1066
Age, Customized [Number; unit: participants]
  <65 years | 540
  >65 and < 75 years | 417
  > 75 years | 109
Sex/Gender, Customized [Number; unit: participants]
  Male | 1066
  Female | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1060
  Black | 3
  Asian | 2
  Other | 1
Total International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms, based on answers to 7questions concerning urinary symptoms: • Incomplete emptying of the bladder • Intermittency • Weak stream • Hesitancy • Frequency • Urgency • Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom. Total score can range from 0 to 35 (mildly symptomatic to severely symptomatic).
  units on a scale | 18.7 (4.41)
Total International Prostate Symptom Score (IPSS) voiding score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 voiding questions (incomplete emptying of the bladder, intermittency, weak stream, hesitancy) and ranges from 0 to 20 (mildly symptomatic to severely symptomatic).
  units on a scale | 9.8 (3.58)
Total International Prostate Symptom Score (IPSS) storage score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires.The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 storage questions (frequency, urgency and nocturia) and ranges from 0 to 15 (mildly symptomatic to severely symptomatic).
  units on a scale | 8.9 (2.37)
IPSS Quality of Life Score(Qol) score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The answers ranged from 0 to 6 (delighted to terrible).
  units on a scale | 4.1 (1.09)
Total Urgency Frequency Score (TUFS) (previous known as Total Urgency Score (TUS) [Mean (Standard Deviation); unit: units on a scale] — FAS population.The Participant Perception of the Intensity of Urgency Scale (PPIUS) is a validated scale completed as part of the micturition diary. For each micturition and/or incontinence episode, the participant rated the degree of associated urgency according to the following 5-point categorical scale: 0.No urgency; 1.Mild urgency; 2.Moderate urgency; 3.Severe urgency; 4.Urgency incontinence. TUFS/TUS was the sum of the PPIUS gradings from the 3-day diary divided by the number of days on which urgency grading was recorded.
  units on a scale | 27.18 (8.59)
Micturitions/24 hour [Mean (Standard Deviation); unit: micturitions] — FAS population. A micturition is any voluntary urination, excluding episodes of incontinence only. The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  micturitions | 11.44 (2.61)
Volume voided/micturition [Mean (Standard Deviation); unit: ml] — FAS population. A micturition is any voluntary urination, excluding episodes of incontinence only. The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  ml | 162.81 (47.57)
Incontinence episodes/24 hour [Mean (Standard Deviation); unit: incontinence episodes] — FAS population. An incontinence episode is defined as an episode with any involuntary loss of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  incontinence episodes | 1.77 (2.04)
Urgency incontinence episodes /24 hour [Mean (Standard Deviation); unit: urgency incontinence episodes] — FAS population. An urgency incontinence episode is defined as an episode with any involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes with PPIUS grade 3 (Severe urgency) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  urgency incontinence episodes | 1.74 (1.97)
Nocturia episodes/ 24 hour [Mean (Standard Deviation); unit: nocturia episodes] — FAS population. A nocturia episode is defined as waking up at night to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  nocturia episodes | 2.40 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety is monitored by collecting AEs, which include abnormal lab parameters, vital signs or ECG data if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study drug or was clinically significant. A serious AE (SAE) was an AE resulting in death, persistent or significant disability/incapacity or congenital anomaly/birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs were assessed by the Investigator for intensity (mild-no disruption of normal daily activities, moderate-affected normal daily activities or severe-inability to perform daily activities) and for causal relationship to study drug. A treatment-emergent adverse event (TEAE) was defined as an AE that occurred after the intake of first dose of double-blind study drug (if on FDC in 905-CL-055) or after first open-label dose until 30 days after the last dose of open-label study drug (in 905-CL-057).
Time Frame: From first dose of double-blind study drug (if on FDC in 905-CL-055) or first open-label dose up to 30 days after last dose of open-label study drug (in 905-CL-057) (up to 56 weeks)
Population: Safety analysis set-participants who received at least 1 dose of the FDC tamsulosin/solifenacin 0.4 mg/6 mg or 0.4 mg/9 mg during the open-label treatment period and had any data reported after the first dose of the FDC during the open-label treatment period
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1066
participants
  Participants With Treatment-Emergent Adverse Event | 499
  Drug-related AEs | 255
  Drug-related SAEs | 12
  Any TEAE causing discontinuation of study drug. | 69

2. Primary Outcome: Change From Baseline to End of Treatment in Post Void Residual (PVR) Volume
Description: PVR volume is the volume of urine retained after voiding. PVR volume was assessed by ultrasonography or bladder scan.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: SAF population with at least one baseline and one post-baseline PVR volume measured.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Total Group
Number analyzed (Participants) | 1056
ml | 10.7 (49.28)

3. Primary Outcome: Change From Baseline to End of Treatment in Maximum Flow Rate (Qmax)
Description: Qmax during a micturition (urination) was recorded using uroflowmetry.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: SAF population with at least one baseine and one post-baseline micturition episode.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Total Group
Number analyzed (Participants) | 1047
ml/s | 4.54 (5.927)

4. Primary Outcome: Change From Baseline to End of Treatment in Average Flow Rate (Qmean)
Description: Qmean during a micturition (urination) was recorded using uroflowmetry.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: SAF population with at least one baseline and one post-baseline micturition episode.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Total Group
Number analyzed (Participants) | 1047
ml/s | 2.05 (2.884)

5. Primary Outcome: Change From Baseline to End of Treatment in Total International Prostate Symptom Score (IPSS)
Description: The International Prostate Symptom Score (IPSS) is a validated global questionnaire to assess the degree of urinary symptoms, based on answers to 7 questions concerning urinary symptoms: • Incomplete emptying of the bladder • Intermittency • Weak stream • Hesitancy • Frequency • Urgency • Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom. Total score can range from 0 to 35 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: Full Analysis Set (FAS)-participants who took at least 1 dose of the FDC during the open-label study, had a total IPSS or TUS at baseline and had at least one total IPSS or TUS after first dose of the FDC in Study 905-CL-057. Excluded 5 participants with invalid questionnaires. Last Observation Carried Forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Group: Participants who received the open-label FDC treatment and were included in the Full Analysis Set of 905-CL-057
Arm/Group | Total Group
Number analyzed (Participants) | 1004
units on a scale | -9.0 (5.69)

6. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Micturitions Per 24 Hours
Description: A micturition is any voluntary urination, excluding episodes of incontinence only.The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Total Group
Number analyzed (Participants) | 1008
micturitions | -2.5 (2.37)

7. Secondary Outcome: Change From Baseline to End of Treatment in Mean Voided Volume Per Micturition
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Total Group
Number analyzed (Participants) | 1008
ml | 39.0 (47.32)

8. Secondary Outcome: Change From Baseline to End of Treatment in Maximum Volume Voided Per Micturition
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The maximum volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Total Group
Number analyzed (Participants) | 1008
ml | 16.6 (101.24)

9. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Urgency Episodes (PPIUS Grade 3 or 4) Per 24 Hours
Description: An urgency episode is defined as an episode of strong desire to void accompanied by fear of leakage or pain. The mean number of urgency episodes with PPIUS grade 3 (Severe urgency) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with at least 1 urgency episode at baseline. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: urgency episodes
Arm/Group | Total Group
Number analyzed (Participants) | 1006
urgency episodes | -3.1 (3.45)

10. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode is defined as an episode with any involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes with PPIUS grade 3 (Severe incontinence) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population and at least 1 urgency incontinence episode at baseline. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: urgency incontinence episodes
Arm/Group | Total Group
Number analyzed (Participants) | 234
urgency incontinence episodes | -1.5 (2.02)

11. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode is defined as an episode with any involuntary loss of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population and at least 1 incontinence episode at baseline. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: incontinence episodes
Groups:
- Total Group: Participants who received the open-label FDC treatment and were included in the Full Analysis Set of 905-CL-057).
Arm/Group | Total Group
Number analyzed (Participants) | 250
incontinence episodes | -1.4 (2.09)

12. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Nocturia Episodes Per 24 Hours
Description: A nocturia episode is defined as waking up at night to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population and at least 1 nocturia episode at baseline. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: nocturia episodes
Arm/Group | Total Group
Number analyzed (Participants) | 968
nocturia episodes | -0.7 (1.05)

13. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Pads Used Per 24 Hours
Description: The mean number of pads per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population and at least 1 use of a pad at baseline. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: pads
Arm/Group | Total Group
Number analyzed (Participants) | 95
pads | -0.9 (1.48)

14. Primary Outcome: Change From Baseline to End of Treatment in Total Urgency Frequency Score (TUFS) (Previously Known as Total Urgency Score [TUS])
Description: The Patient Perception of the Intensity of Urgency Scale (PPIUS) is a validated scale completed as part of the micturition diary. For each micturition and/or incontinence episode, the participant rated the degree of associated urgency according to the following 5-point categorical scale: • 0. No urgency; • 1. Mild urgency; • 2. Moderate urgency; • 3. Severe urgency; • 4. Urgency incontinence TUS/TUFS was calculated as the sum of the PPIUS gradings from the 3-day diary divided by the number of days on which urgency grading was recorded. Higher scores indicate more severe urgency.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1005
units on a scale | -10.1 (9.23)

15. Secondary Outcome: Change From Baseline to End of Treatment in IPSS Voiding Score
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 voiding questions (incomplete emptying of the bladder, intermittency, weak stream, hesitancy) and ranges from 0 to 20 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: A total of 5 subjects has been excluded from the FAS analysis due to invalid questionnaires. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1004
units on a scale | -4.7 (4.09)

16. Secondary Outcome: Change From Baseline to End of Treatment in IPSS Storage Score
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms based on answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 storage questions (frequency,urgency and nocturia) and ranges from 0 to 15 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: A total of 5 subjects has been excluded from the FAS analysis due to invalid questionnaires. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1004
units on a scale | -4.3 (2.88)

17. Secondary Outcome: Change From Baseline to End of Treatment in IPSS Quality of Life (QoL) Score
Description: The QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The answers ranged from 0 to 6 (delighted to terrible).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: FAS population with data available at both baseline and end of treatment and the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1003
units on a scale | -1.9 (1.53)

18. Secondary Outcome: Change From Baseline to End of Treatment in Individual IPSS Scores
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms, based on answers to 7 questions concerning urinary symptoms: • Incomplete emptying of the bladder • Intermittency • Weak stream • Hesitancy • Frequency • Urgency • Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: A total of 5 subjects has been excluded from the FAS analysis due to invalid questionnaires. LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1004
units on a scale
  Incomplete emptying of the bladder | -1.3 (1.49)
  Frequency | -1.7 (1.41)
  Intermittency | -1.0 (1.48)
  Urgency | -1.8 (1.54)
  Weak stream | -1.6 (1.62)
  Hesitancy | -0.8 (1.42)
  Nocturia | -0.9 (1.17)

19. Secondary Outcome: Change From Baseline to End of Treatment in Symptom Bother Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The Symptom Bother portion consists of an 8-item scale scored from 1 to 6.The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1003
units on a scale | -20.6 (17.45)

20. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQoL) Subscale: Coping Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: • coping • concern • sleep • social interaction Coping score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1000
units on a scale | 17.3 (18.98)

21. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQoL) Subscale: Concern Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: • coping • concern • sleep • social interaction Concern score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1000
units on a scale | 15.0 (18.15)

22. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQoL) Subscale: Sleep Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: • coping • concern • sleep • social interaction Sleep score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1001
units on a scale | 15.3 (19.61)

23. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQoL) Subscale: Social Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: • coping • concern • sleep • social interaction Social score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1002
units on a scale | 7.6 (15.15)

24. Secondary Outcome: Change From Baseline to End of Treatment in Health-related Quality of Life (HRQoL) Subscale: Total Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: • coping • concern • sleep • social interaction Total score is calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1000
units on a scale | 14.3 (15.59)

25. Secondary Outcome: Number of OAB-q Responders Based on Health-related Quality of Life: Total Score
Description: A OAB-q responder was defined as a participant with an improvement from baseline in HRQoL subscale total score ≥ 10.
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Total Group
Number analyzed (Participants) | 1000
percentage of participants | 55.7

26. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Mobility Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: • mobility • self-care • usual activity • pain/discomfort • anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = confined to bed).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1003
participants
  No problem -> No problem | 775
  No problem -> Some problem | 58
  No problem -> confined to bed | 1
  No problem -> no data | 0
  Some problem -> No problem | 67
  Some problem -> Some problem | 102
  Some problem -> confined to bed | 0
  Some problem -> No data | 0
  Confined to bed -> no problem | 0
  Confined to bed -> some problem | 0
  Confined to bed -> confined to bed | 0
  Confined to bed -> no data | 0
  No data -> no problem | 1
  No data -> some problem | 0
  No data -> confined to bed | 0
  No data -> no data | 0

27. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Self-care Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: • mobility • self-care • usual activity • pain/discomfort • anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = unable to wash/dress).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1001
participants
  No problem -> No problem | 934
  No problem -> Some problem | 27
  No problem -> Unable to wash/dress | 1
  No problem -> No data | 0
  Some problem -> no problem | 18
  Some problem -> some problem | 19
  Some problem -> unable to wash/dress | 0
  Some problem -> no data | 0
  Unable to wash/dress -> no problem | 2
  Unable to wash/dress -> some problem | 0
  Unable to wash/dress -> unable to wash/dress | 0
  Unable to wash/dress -> no data | 0
  No data -> no problem | 3
  No data -> some problem | 0
  No data -> unable to wash/dress | 0
  No data -> no data | 0

28. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Usual Activities Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: • mobility • self-care • usual activity • pain/discomfort • anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = unable to perform usual activities).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1003
participants
  No problem -> No problem | 805
  No problem -> Some problem | 54
  No problem -> unable to perform usual activities | 1
  No problem -> no data | 0
  Some problem -> no problem | 80
  Some problem -> some problem | 60
  Some problem -> unable to perform usual activities | 0
  Some problem -> no data | 0
  Unable to perform usual activities -> no problem | 1
  Unable to perform usual activities -> some problem | 2
  Unable to perform usual activities -> same status | 0
  Unable to perform usual activities -> no data | 0
  No data -> no problem | 1
  No data -> some problem | 0
  No data -> unable to perform usual activities | 0
  No data -> no data | 0

29. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Pain/Discomfort Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: • mobility • self-care • usual activity • pain/discomfort • anxiety/depression Each domain has 3 response levels (1= no pain, 2= moderate pain, 3 = extreme pain).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1002
participants
  No pain -> no pain | 499
  No pain -> moderate pain | 71
  No pain -> extreme pain | 2
  No pain -> no data | 0
  Moderate pain -> no pain | 202
  Moderate pain -> moderate pain | 200
  Moderate pain -> extreme pain | 5
  Moderate pain -> no data | 0
  Extreme pain -> no pain | 10
  Extreme pain -> moderate pain | 7
  Extreme pain -> extreme pain | 6
  Extreme pain -> no data | 0
  No data -> no pain | 2
  No data -> moderate pain | 0
  No data -> extreme pain | 0
  No data -> no data | 0

30. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Anxiety/Depression Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: • mobility • self-care • usual activity • pain/discomfort • anxiety/depression Each domain has 3 response levels (1= not anxious, 2= moderately anxious, 3 = extremely anxious).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Total Group
Number analyzed (Participants) | 1003
participants
  Not anxious -> Not anxious | 737
  Not anxious -> moderately anxious | 37
  Not anxious -> extremely anxious | 1
  Not anxious -> no data | 0
  Moderately anxious -> not anxious | 103
  Moderately anxious -> moderately anxious | 109
  Moderately anxious -> extremely anxious | 3
  Moderately anxious -> no data | 0
  Extremely anxious -> not anxious | 4
  Extremely anxious -> moderately anxious | 4
  Extremely anxious -> extremely anxious | 5
  Extremely anxious -> no data | 0
  No data -> not anxious | 1
  No data -> moderately anxious | 0
  No data -> extremely anxious | 0
  No data -> no data | 0

31. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Visual Analogue Scale (VAS) Score
Description: Visual Analogue Scale (VAS) is part of the EQ-5D questionnaire. The VAS is self-rated by the participant ranging from 0 to 100 (worst imaginable health state to best imaginable health state).
Time Frame: Baseline and up to 52 weeks of FDC treatment
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Group
Number analyzed (Participants) | 1000
units on a scale | 6.4 (17.15)

ADVERSE EVENTS:
Time Frame: From first dose of double-blind study drug (if on FDC in 905-CL-055) or first open-label dose up to 30 days after last dose of open-label study drug (in 905-CL-057) (up to 56 weeks)
Arm/Group | Total Group
Serious Adverse Events (participants affected / at risk) | 64/1066
Other Adverse Events (participants affected / at risk) | 180/1066
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Group (N=1066)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Cerebral disorder (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Lateral medullary syndrome (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 6
Renal failure acute (Renal and urinary disorders) | 2
Calculus ureteric (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchietasis (Infections and infestations) | 1
Lobar pnemonia (Infections and infestations) | 1
Aortic aneurysm (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Femoral arterial stenosis (Vascular disorders) | 1
Iliac artery occulsion (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Cataract (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Group (N=1066)
Constipation (Gastrointestinal disorders) | 55 (61)
Dry Mouth (Gastrointestinal disorders) | 132 (138)

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principle Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 90 days prior to publication for review and comment. Sponsor may delay the publication to seek patent approval.